CLINICAL TRIAL: NCT06063213
Title: Using Transcriptional Assessment of Immune Response to Assess Immunosuppression After Liver Transplantation
Acronym: TGI
Status: Active, not recruiting | Type: Observational
Sponsor: University of Florida (Other)
Collaborators: Transplant Genomics, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: IRB202300021
Record Dates: First submitted 2023-09-26; First posted 2023-10-02 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2025-01

CONDITIONS: Transplant Complication

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Liver Transplant Group: Patients <1 month post-surgery for liver transplant only.
- Liver-Kidney Transplant Group: Patients <1 month post-surgery for simultaneous kidney-liver transplant only.

SUMMARY:
To develop a prospective quantitative liver allograft monitoring protocol and retrospectively validate the use of Phenotypic personalized medicine (PPM) in immunosuppression dosing in liver transplant recipients.

DETAILED DESCRIPTION:
The investigators have developed a computational approach, Phenotypic Personalized Medicine (PPM), to utilize empiric clinical data to construct patient-specific visual maps that represent each individual's phenotypic response to drug treatment. Because this process does not require a priori knowledge of disease mechanism, it can effectively personalize drug dosing for any disease despite frequent changes to treatment regimens or patient physiology and genetics. In a pilot randomized controlled trial and its follow-up larger trial, the investigators have shown that transplant patients prospectively dosed with PPM-determined tacrolimus doses had improved drug trough-level management compared with standard of care physician-determined tacrolimus doses.

The ultimate objective in this project is to improve graft and patient outcomes in solid organ transplant recipients by using PPM to optimize immunosuppression dosing. The investigators hypothesize that existing and clinically validated quantifiable markers of immune state and allograft injury are clinically useful measures that can be employed with PPM as actionable analytical inputs for a dynamic optimization of patient-specific immunosuppression. The investigators will test this hypothesis by developing a prospective quantitative liver allograft monitoring protocol and validate the use of PPM in immunosuppression dosing in liver transplant recipients.

This study constitutes the first step in developing and then validating a personalized immunosuppression platform. The mechanism-independent nature of PPM ensures that it will be adaptive and actionable so that it can be applied to diverse sets of patients. The scalability of PPM also ensures that it can be deployed at a scale that can be applied widely to patients receiving care regardless of location.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age
* At least one-month post-transplant
* Recipient of a liver transplant alone or a simultaneous liver-kidney transplant

Exclusion Criteria:

* Unwilling to provide informed consent
* Recipient of a previous bone marrow or stem cell transplant
* Pregnant
* Unlikely to be able to comply with the study requirements, as determined by the PI

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients that are simultaneous Liver Kidney Transplant recipients that are one month post transplant. Patients that are Liver Transplant recipients that are one month post transplant.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2023-12-15 (Actual); Primary Completion 2026-10-15 (Estimated); Study Completion 2026-10-15 (Estimated)

PRIMARY OUTCOMES:
Episodes of rejection | 6 months
  Patients will be followed for six months after transplantation according to standard of care. Episodes of biopsy proven rejection will be counted.

SECONDARY OUTCOMES:
Episodes of infection | 6 months
  Patients will be followed for six months after transplantation according to standard of care. Episodes of culture positive infection will be counted.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Florida, Gainesville, Florida, United States